CLINICAL TRIAL: NCT02138721
Title: Local Treatment With Radical Prostatectomy (RP) for Newly-diagnosed Metastatic Prostate Cancer (mPCa).
Brief Title: Local Treatment With RP for Newly-diagnosed mPCa
Acronym: LoMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B670201420709
Record Dates: First submitted 2014-05-08; First posted 2014-05-15 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Prostatic Neoplasms; Neoplasm Metastasis
Keywords: Metastatic Prostate Cancer; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No local treatment (No Intervention): Routine care in metastatic prostate cancer.
- Local treatment (Experimental): Radical Prostatectomy (RP) + routine care in metastatic prostate cancer.
  Interventions: Procedure: Radical Prostatectomy (RP)

INTERVENTIONS:
Procedure: Radical Prostatectomy (RP) — Radical Prostatectomy with extended Pelvic Lymph Node Dissection within 8 weeks after inclusion.
  Arms: Local treatment

SUMMARY:
The objective of this study is to evaluate the role of local treatment with radical prostatectomy in patients with newly-diagnosed metastatic hormone-sensitive prostate cancer.

DETAILED DESCRIPTION:
Patients recently diagnosed with metastatic prostate cancer (mPCa), and meeting the eligibility criteria, will be given the opportunity to enroll in this study.

Study Groups:

After inclusion, patients requesting local treatment can undergo radical prostatectomy (RP) with pelvic lymph-node dissection (PLND) after multi-disciplinary evaluation. This resulting in a local treatment group and a no local treatment group. For ethical reasons, no randomization will be done.

Follow-up:

Patients not undergoing local treatment will undergo the current standard of care in our institution. And besides the intervention of local treatment, the other patients will receive this same current standard of care.

Routine follow-up visits, with physical examination, laboratory tests and questionnaires, will be scheduled every 3 months. A CT-scan (abdomen-pelvis) and bone scan will be performed if a clinical progression is diagnosed or suspected and when Castration Refractory PCa (CRPC) is established.

Androgen Deprivation Therapy (ADT) will be initiated in case of one of the following:

* symptoms related to metastatic lesion(s)
* Prostate Specific Antigen (PSA) > 50ng/ml and doubling time (PSA-DT) < 6 months (starting 3 months after inclusion at earliest)

The estimated number of patients to be included in the local treatment arm is 40.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate adenocarcinoma, confirmed by histology
* Newly diagnosis of metastatic disease (stage TanyNanyM+)
* Life expectancy ≥2y based on comorbid conditions, WHO performance status 0-2
* Written informed consent, male ≥18yo
* Willing and expected to comply with study protocol and follow-up schedule
* Multidisciplinary Oncologic Consultation (MOC) approval

Exclusion Criteria:

* Previous local or systemic treatment for prostate cancer
* Metastatic brain disease, leptomeningeal disease or imminent spinal cord compression
* Symptoms clearly related to metastatic lesions
* Any other previous or current (malignant) disease which, in the judgment of the responsible physician, is likely to interfere with LoMP treatment or assessment

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Castration Refractory Prostate Cancer Progression-Free Survival | up to 10 years
  From date of inclusion until the date of Castration Refractory Prostate Cancer (CRPC) defined according to European Association of Urology (EAU) guidelines, or date of death from any cause, whichever came first, assessed up to 10 years. [months]
Time to first Disease Related Event | up to 10 years
  From date of inclusion until the date of any event related to local disease progression (eg ureter obstruction, bladder outlet obstruction), any Skeletal Related Event (SRE) or any event related to metastasis (eg lymphedema). [months]

SECONDARY OUTCOMES:
Overall Survival | at year 1 - 2 - 5
  From date of inclusion until the date of death from any cause, assessed up to 10 years. [months]
Prostate Cancer Specific Survival | at year 1 - 2 - 5
  From date of inclusion until the date of death due to prostate cancer, assessed up to 10 years. [months]
Quality of Life | at month 6 - 12
  Evaluated by the EuroQoL 5 Dimensions 5 Levels Questionnaire
Time to Androgen Deprivation Therapy start | up to 10 years, estimated to occur within 24 months
  From date of inclusion until the date of start of Androgen Deprivation Therapy (ADT) (criteria described in protocol) [months]

OTHER OUTCOMES:
Cytoreductive effect of local treatment in metastatic disease lesions [%] | at month 3 - 6
  Tumor burden assessment will be performed by image-based evaluation (RECIST criteria v1.1) when possible.
Cost-effectiveness of local treatment arm versus no local treatment arm | analysis after trial ending, estimated in 10-15 years
  Evaluation of cost [€] and quality-adjusted life years [QALYs] related to interventions needed in both arms from inclusion to death.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Lumen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (5):
- Belgium (5):
  - ASZ Aalst, Aalst
  - Imelda Ziekenhuis, Bonheiden
  - University Hospital, Ghent, Ghent
  - Sint-Fransiskusziekenhuis, Heusden-Zolder
  - AZ Jan Portaels, Vilvoorde

REFERENCES:
- [Result] Poelaert F, Verbaeys C, Rappe B, Kimpe B, Billiet I, Plancke H, Decaestecker K, Fonteyne V, Buelens S, Lumen N. Cytoreductive Prostatectomy for Metastatic Prostate Cancer: First Lessons Learned From the Multicentric Prospective Local Treatment of Metastatic Prostate Cancer (LoMP) Trial. Urology. 2017 Aug;106:146-152. doi: 10.1016/j.urology.2017.02.051. Epub 2017 Apr 20. PMID 28435034